CLINICAL TRIAL: NCT05050461
Title: Immune Response After SARS-CoV-2 Vaccination in a Context of Non-Hodgkin Lymphoma
Brief Title: Immune Response After SARS-CoV-2 (COVID-19) Vaccination in a Context of Non-Hodgkin Lymphoma
Acronym: LYMPHO-CoVac
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Given the evolution of Covid 19, patient inclusions became very difficult or even non-existent in all participating centers over time
Sponsor: Versailles Hospital (Other)
Responsible Party: Principal Investigator, Caroline BESSON, Investigator Coordinator, Versailles Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: P21/08 - LYMPHO-CoVac
Record Dates: First submitted 2021-09-13; First posted 2021-09-20 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Non-hodgkin Lymphoma,B Cell; Vaccination Failure

STUDY DESIGN:
Intervention Model Description: There will be an arm foses and an arm for controls
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cases (Active Comparator): Patients with a history of B-NHL
  Interventions: Other: Immunological analyses
- Controls (Other): Spouses of cases
  Interventions: Other: Immunological analyses

INTERVENTIONS:
Other: Immunological analyses — Immunological analyses will be performed at inclusion in both arms

SUMMARY:
The specific immune response to SARS-CoV-2 includes a humoral response - specific IgM appearing 5 days after the onset of symptoms while IgG appears after 14 days - and a T lymphocyte component, with specific activated CD8 and CD4 T lymphocytes.

Mortality from infection varies greatly depending on the age of the affected subjects and their comorbidities including a history of cancer. Among these cancers, a history of malignant hemopathy in the 5 years preceding the onset of Covid-19 increases the risk of death by a factor of 3. Among them, lymphoid hemopathies induce hypogammaglobulinemia and / or lymphopenia. These factors combined with chemotherapy and immunotherapy treatments promote the development of infections in affected individuals. Among these, are the anti-CD20 monoclonal antibodies, widely prescribed for treating B-cell non-Hodgkin lymphomas (B-NHL). They induce a deep and lasting B-cell lymphopenia, which can promote infections. They reduce the production of antibodies and the constitution of memory responses to a new pathogen or to a vaccination. In addition, B lymphocytes likely have a key immunomodulatory role in the control of viral infections.

A retrospective study in 89 patients with lymphoma and Covid-19 were conducted after the first phase of the epidemic in different centers in the Île-de-France and eastern France regions. With a 6-month follow-up, a pejorative prognostic impact of anti-CD20 monoclonal antibody treatment on Covid-19-related mortality were showed.

Vaccination of these at-risk patients is therefore essential. A growing concern is how patients with B-NHL who have been vaccinated with a SARS-CoV-2 mRNA vaccine are protected against infection, depending on whether or not they have received anti-CD20 monoclonal drugs and / or chemotherapy.

Knowing the medium-term immunological evolution after vaccination against SARS-CoV-2 in patients with B-cell NHL is necessary in order to be able to adapt the therapeutic and vaccine recommendations.

The main objective of this study is to determine how recent treatment (in the year before vaccination) with anti-CD20 monoclonal antibody modifies the immune response after vaccination against SARS-CoV-2 in adults with B-NHL compared to patients who have not recently been exposed to this immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Adult aged at least 18 years old

  * Having received (at least) two injections of anti-SARS-CoV-2 messenger RNA vaccine (Pfizer and / or Moderna)
  * Affiliated to social security
  * consenting to the study
  * Concerning cases only: Be or have been affected by B-NHL in remission, active surveillance or during first-line or second-line treatment, regardless of this treatment

Exclusion Criteria:

Patient less than 18 years old

* Patient with protective measure (curatorship, guardianship, safeguard of justice, deprived of liberty, in an emergency situation)
* Patient unable to express their consent
* Pregnant or breastfeeding woman
* Patient refusing to participate
* Concerning cases: Patient whose life expectancy related to B-NHL is less than 6 months, History of allogeneic hematopoietic stem cell transplantation, Patient with CART cells treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
Comparison of humoral (especially anti-SARS-CoV-2 antibody levels) and T cell memory responses in adult patients with B-NHL depending on whether or not they were exposed to anti-CD20 monoclonal antibody treatment in the year before vaccination. | at inclusion

CONTACTS AND LOCATIONS:
Locations (7):
- France (7):
  - Emile Muller Hospital, Hematology unit, Mulhouse
  - Institut of Cancerology Strasbourg Europe (ICANS), Hematology deparment, Strasbourg
  - Hospitals of Brabois, Hematology unit, Vandœuvre-lès-Nancy
  - André Mignot -Versailles Hospital, Hemato-oncology unit, Le Chesnay, Île-de-France Region
  - saint Louis Hospital, Hemato-oncology unit, Paris, Île-de-France Region
  - Saint Antoine Hospital, Hematology unit, Paris, Île-de-France Region
  - Pitié Salpêtrière Hospital, Hematology unit, Paris, Île-de-France Region

REFERENCES:
- [Background] Dan JM, Mateus J, Kato Y, Hastie KM, Yu ED, Faliti CE, Grifoni A, Ramirez SI, Haupt S, Frazier A, Nakao C, Rayaprolu V, Rawlings SA, Peters B, Krammer F, Simon V, Saphire EO, Smith DM, Weiskopf D, Sette A, Crotty S. Immunological memory to SARS-CoV-2 assessed for up to 8 months after infection. Science. 2021 Feb 5;371(6529):eabf4063. doi: 10.1126/science.abf4063. Epub 2021 Jan 6. PMID 33408181
- [Background] Liang W, Guan W, Chen R, Wang W, Li J, Xu K, Li C, Ai Q, Lu W, Liang H, Li S, He J. Cancer patients in SARS-CoV-2 infection: a nationwide analysis in China. Lancet Oncol. 2020 Mar;21(3):335-337. doi: 10.1016/S1470-2045(20)30096-6. Epub 2020 Feb 14. No abstract available. PMID 32066541
- [Background] Maschmeyer G, De Greef J, Mellinghoff SC, Nosari A, Thiebaut-Bertrand A, Bergeron A, Franquet T, Blijlevens NMA, Maertens JA; European Conference on Infections in Leukemia (ECIL). Infections associated with immunotherapeutic and molecular targeted agents in hematology and oncology. A position paper by the European Conference on Infections in Leukemia (ECIL). Leukemia. 2019 Apr;33(4):844-862. doi: 10.1038/s41375-019-0388-x. Epub 2019 Jan 30. PMID 30700842
- [Background] Lamure S, Dulery R, Di Blasi R, Chauchet A, Laureana C, Deau-Fischer B, Drenou B, Soussain C, Rossi C, Noel N, Choquet S, Bologna S, Joly B, Kohn M, Malak S, Fouquet G, Daguindau E, Bernard S, Thieblemont C, Cartron G, Lacombe K, Besson C. Determinants of outcome in Covid-19 hospitalized patients with lymphoma: A retrospective multicentric cohort study. EClinicalMedicine. 2020 Oct;27:100549. doi: 10.1016/j.eclinm.2020.100549. Epub 2020 Oct 13. PMID 33073216
- [Background] Dulery R, Lamure S, Delord M, Di Blasi R, Chauchet A, Hueso T, Rossi C, Drenou B, Deau Fischer B, Soussain C, Feugier P, Noel N, Choquet S, Bologna S, Joly B, Philippe L, Kohn M, Malak S, Fouquet G, Daguindau E, Taoufik Y, Lacombe K, Cartron G, Thieblemont C, Besson C. Prolonged in-hospital stay and higher mortality after Covid-19 among patients with non-Hodgkin lymphoma treated with B-cell depleting immunotherapy. Am J Hematol. 2021 Aug 1;96(8):934-944. doi: 10.1002/ajh.26209. Epub 2021 May 12. PMID 33909916